CLINICAL TRIAL: NCT05468216
Title: The Effect of MovIn-Lessons Project on Physical Activity Levels, Executive Functions, Academic Performance and On-task Behaviour in Primary Schools: Study Protocol for a Cluster-randomized Controlled Trial
Brief Title: Movement Integration in Primary Schools' Lessons
Acronym: MovIn-Lessons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Anna M. Señé Mir, PhD, Lecturer and researcher, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MovIn
Record Dates: First submitted 2022-05-09; First posted 2022-07-21 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Physical Activity; Executive Function
Keywords: exercise; education; sedentary behaviour; movement integration; executive functions; academic performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Only an allocation concealment mechanism will be used to prevent clusters' selection bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MovIn-Lessons group (Experimental): The schools which will implement the movement integration in the learning activities of primary education subjects (maths, natural science and English).
  Interventions: Other: MovIn-Lessons group
- Control group (No Intervention): Schools which will continues applying the same methodology in the realization of the learning activities.

INTERVENTIONS:
Other: MovIn-Lessons group — The MovIn-Lessons intervention will consist of infusing PA in math, English and natural sciences lessons in primary education. The movement will be integrated in the learning activities for at least 20 minutes per session, at different physical intensities.
  Arms: MovIn-Lessons group

SUMMARY:
The study assesses the effects of long-term movement integration intervention in academic lessons of primary education (6th grade) on physical activity levels and sedentary behaviour, executive functions, academic achievement and on-task behaviour. To achieve it, a cluster randomized controlled trial design will be adopted, where schools will be the clusters.

DETAILED DESCRIPTION:
The evidence shows that over 50% of Spanish children do not achieve the PA recommendations established by the WHO, and are therefore at higher risk of both short-term (e.g., overweight and obesity) and long-term health consequences (chronic illness in adolescence and adulthood). This is an alarming social and public health challenge in Spain and across Europe and effective solutions are needed.

Therefore, in this cluster randomized controlled trial, it will be tested if a long-term movement integration intervention in academic lessons (MovIn-Lessons) in primary education (specifically 6th grade) can increase the physical activity levels of children and reduce the sedentary behaviour at school-time. Additionally, it will be tested if this intervention can improve the executive functions, academic achievement and on-task behaviour.

Movement integration is defined as infusing physical activity, at any level of intensity, within general education classrooms during school time. Specifically, MovIn-Lessons intervention will consist of infusing physical activity in math, English and natural sciences lessons for all children attending the intervention schools. This will be achieved by carrying out learning activities in an active way.

Participants include children that are studying the 6th grade in primary education schools. Due to the cluster-randomized controlled trial design, the schools will be the clusters, and the design will have a restriction. The restriction is each cluster (school) that participates has to be from different towns or cities, even if schools are allocated to the same arm (intervention or control group). The aim of this restriction is to preserve construct validity by avoiding the fact that children from different schools in the same town or city could communicate with each other.

The recruitment will be following this procedure: all Catalan schools in the provinces of Barcelona and Girona will receive an invitation to participate in the study. Schools that are interested in taking part and meet the inclusion criteria will be eligible to participate. Schools will be randomly allocated to intervention or control group with matching. The matching criteria will be schools' characteristics (public or private, geographic location, sociodemographic profile and number of sixth grade classrooms) and teachers' characteristics (experience, confidence and pedagogical models used). Additionally, an allocation concealment mechanism will be used to prevent clusters' selection bias. All eligible participants will complete baseline assessments and follow-up evaluations conducted in the middle of the intervention (after three months), and one-week post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* children in sixth grade of primary education

Exclusion Criteria:

* children who require special educational needs and it is not following the whole-group classes

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Physical activity measures change: time and intensity | Baseline, 8 weeks after starting intervention, end of the intervention (after 16 weeks)
  Accelerometers will be used to measure and quantify the physical activity levels of students. Accelerometers have already been demonstrated as a valid and objective measure to quantify body posture and activity patterns during free-living conditions in children and adults.
Sedentary behaviour measures change: time | Baseline, 8 weeks after starting intervention, end of the intervention (after 16 weeks).
  Accelerometers will be used to measure and quantify sedentary behaviour of students. Accelerometers have already been demonstrated as a valid and objective measure to quantify body posture and activity patterns during free-living conditions in children and adults.
Executive functions measures change | Baseline, 8 weeks after starting intervention, end of the intervention (after 16 weeks)
  Three core EFs will be assessed with validated tests from the NIH toolbox battery for the population aged between 3 and 85 years old. Inhibition control and attention: Flanker Inhibitory Control and Attention test; Working memory: List Sorting Working Memory test; Cognitive flexibility: Dimensional Change Card Sort test.
Academic achievement measures change | Baseline, and end of the intervention (after 16 weeks)
  The Catalan national standardized test consists of evaluating the degree of achievement of basic competences at the end of primary education (sixth grade).
On-task behaviour measures change | Baseline, 8 weeks after starting intervention, end of the intervention (after 16 weeks)
  The Direct Behaviour Rating Scale assesses students' behaviour and engagement by rating the percentage of time that the student does the desired behaviour. High scores on the Direct Behavior Rating scales (Academically engaged, Respectful and Disruptive) indicate high levels, with 10 being the maximum value. On the other hand, low scores on the Direct Behavior Rating scales (Academically engaged, Respectful and Disruptive) indicate low levels, with 0 being the minimum value.

OTHER OUTCOMES:
Socioeconomic status | Baseline
  (confounding variable) The Family Affluence Scale II (FAS II) consists of four questions asking children aspects they are likely to know about their family. FAS II low (score=0,1,2) indicates low affluence, FAS II medium (score=3,4,5) indicates middle affluence, and FAS II high (score=6,7,8,9) indicates high affluence. Therefore 0 is the minimum value and 9 the maximum value.
General Physical activity levels | Baseline
  (confounding variable) The Physical Activity Questionnaire for Children (PAQ-C) assesses the general physical activity level in the last seven days. It is a self-administered recall questionnaire.
Body Mass Index | Baseline
  (confounding variable)

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Señé Mir, PhD, Principal Investigator — University of Vic- Central University of Vic
Locations (1):
- University of Vic- Central University of Catalonia, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No